CLINICAL TRIAL: NCT05623696
Title: Effect of Repetitive Transcranial Magnetic Stimulation (rTMS) of the Dorsolateral Prefrontal Cortex (DLPFC) on Hypercapnic Air Hunger Induced in Healthy Individuals.
Brief Title: Effect of Non-invasive Magnetic Stimulation of the Brain on Breathlessness in Healthy Individuals.
Acronym: AHrTMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oxford Brookes University (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Dr. Shakeeb H Moosavi, Reader in Clinical Physiology, Oxford Brookes University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HLS/2021/PH/002
Record Dates: First submitted 2022-11-12; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Dyspnea
Keywords: Air Hunger
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Intervention Model Description: Following a practice session, there will be 3 intervention arms presented in random order on 3 separate days. The three arms will be: (i) 10-20mins of 5Hz rTMS over left DLPFC (Arm 1), (ii) 5Hz rTMS over right DLPFC (Arm 2), (iii) sham rTMS (Arm 3). A standard steady state air hunger test will be conducted before and immediately after each intervention.
Who Masked: Participant
Masking Description: Masking will only be applied to the participants in relation to whether they receive sham or actual rTMS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stimulation of Left DLPFC (Experimental): Intervention applied to Left DLPFC located by the BeamF3 technique
  Interventions: Device: Sham or actual non-invasive (Magnetic) brain stimulation
- Stimulation of Right DLPFC (Active Comparator): Intervention applied to Right DLPFC located by the BeamF3 technique
  Interventions: Device: Sham or actual non-invasive (Magnetic) brain stimulation
- Sham Stimulation (Sham Comparator): Sham intervention applied to either the left or right DLPFC
  Interventions: Device: Sham or actual non-invasive (Magnetic) brain stimulation

INTERVENTIONS:
Device: Sham or actual non-invasive (Magnetic) brain stimulation — 5 Hz rTMS applied using an actual or sham coil over the left or right DLPFC
  Other Names: MagStim

SUMMARY:
The purpose of this study is to see if the front part of the brain called the "Dorsolateral Prefrontal Cortex" (DLPFC) has a role in our ability to feel breathlessness. The experiment will use a device that sits on the top of the head which produces a magnetic field that penetrates the scalp and excites the brain tissue directly under it. This procedure is called repetitive transcranial magnetic stimulation (rTMS), it is a painless procedure and known to be safe in healthy individuals. Previous research has shown that the pain felt when capsaicin, the active ingredient in 'chilli' powder, is applied to the hand is reduced by applying the rTMS on the scalp directly above the DLPFC part of the brain. In this experiment we want to see if breathlessness is also reduced. We will use a breathing task that will generate a moderate amount of breathlessness by adding a small amount of carbon dioxide to the inhaled air, while preventing the increase in the amount of breathing we would normally see in response to this. If we find that breathlessness produced by this breathing task is reduced after rTMS over the DLPFC, this may lead to new drugs that target this part of the brain in patients suffering from breathlessness due to heart or lung disease. The study will also improve our knowledge of how the brain enables us to feel breathlessness

ELIGIBILITY:
Inclusion Criteria:

healthy individuals, over 18 years old, with no history of heart, lung or neurological conditions

Exclusion Criteria:

* Any history of respiratory problems (including Asthma that involves regular use of inhalers)
* Any history of heart or circulatory problems (e.g. palpitations, arrhythmias, angina, BP)
* Any history of epilepsy, convulsions or seizures, migraines, or fainting
* Any history of anxiety disorders (e.g. panic attacks)
* Any history of serious head injury or brain surgery
* Any metal parts in the head (except dental wire)
* Any implants (e.g. pacemaker, insulin pump, neurostimulator)
* Pregnancy or problems with alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Air hunger | Average of 4 steady state ratings in the last minute of air hunger tests
  Visual analog scale ratings of air hunger

SECONDARY OUTCOMES:
Mood assessment | immediately following pre and post intervention air hunger tests
  Bond Lader Mood questionnaire
Trait and state anxiety scores | immediately following pre and post intervention air hunger tests
  Spielberger's State-Trait anxiety inventory
Dyspnoea-12 total, physical and emotion scores | Administered immediately following pre and post intervention air hunger tests in relation to the "test just completed"
  Multidimensional D12-Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Shakeeb H Moosavi, PhD, Principal Investigator — Oxford Brookes University
Locations (1):
- Oxford Brookes University, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banzett RB, Moosavi SH. Dyspnea and pain: Similarities and contrasts between two very unpleasant sensations. APS Bulletin. 2001; 11: 1-8.
- [Background] Brighina F, De Tommaso M, Giglia F, Scalia S, Cosentino G, Puma A, Panetta M, Giglia G, Fierro B. Modulation of pain perception by transcranial magnetic stimulation of left prefrontal cortex. J Headache Pain. 2011 Apr;12(2):185-91. doi: 10.1007/s10194-011-0322-8. Epub 2011 Feb 25. PMID 21350791
- [Background] Harrison OK, Hayen A, Wager TD, Pattinson KTS. Investigating the specificity of the neurologic pain signature against breathlessness and finger opposition. Pain. 2021 Dec 1;162(12):2933-2944. doi: 10.1097/j.pain.0000000000002327. PMID 33990110
- [Background] Herigstad M, Hayen A, Evans E, Hardinge FM, Davies RJ, Wiech K, Pattinson KTS. Dyspnea-related cues engage the prefrontal cortex: evidence from functional brain imaging in COPD. Chest. 2015 Oct;148(4):953-961. doi: 10.1378/chest.15-0416. PMID 26134891
- [Background] Nierat MC, Hudson AL, Chaskalovic J, Similowski T, Laviolette L. Repetitive transcranial magnetic stimulation over the supplementary motor area modifies breathing pattern in response to inspiratory loading in normal humans. Front Physiol. 2015 Sep 29;6:273. doi: 10.3389/fphys.2015.00273. eCollection 2015. PMID 26483701
- [Background] Yorke J, Moosavi SH, Shuldham C, Jones PW. Quantification of dyspnoea using descriptors: development and initial testing of the Dyspnoea-12. Thorax. 2010 Jan;65(1):21-6. doi: 10.1136/thx.2009.118521. Epub 2009 Dec 8. PMID 19996336